CLINICAL TRIAL: NCT00114790
Title: Boronophenylalanine (BPA)-Based Boron Neutron Capture Therapy (BNCT) in the Treatment of Inoperable and Irradiated Head and Neck Tumors: A Feasibility Study
Brief Title: Boronophenylalanine (BPA)-Based Boron Neutron Capture Therapy (BNCT) in the Treatment Head and Neck Tumors
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Boneca Corporation (Industry)
Responsible Party: Principal Investigator, Professor Heikki Joensuu, professor, Helsinki University Central Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HN-BPA-01-2003
Record Dates: First submitted 2005-06-17; First posted 2005-06-20 (Estimated); Last update posted 2013-05-06 (Estimated); Status verified 2013-05

CONDITIONS: Head and Neck Cancer
Keywords: head and neck cancer; boron neutron capture therapy; radiation therapy; boronophenylalanine
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BNCT. (Experimental): Boronophenylalanine-based BNCT.
  Interventions: Radiation: boronophenylalanine-based BNCT

INTERVENTIONS:
Radiation: boronophenylalanine-based BNCT — Boronophenylalanine is infused into a peripheral vein prior to neutron irradiation.

SUMMARY:
Boron Neutron Capture Therapy (BNCT) is an experimental radiation therapy technique which is based on the principle of irradiating boron atoms with neutrons. When neutrons have relatively low energy, boron atoms that have been targeted to cancerous tissue using a suitable boron carrier (an amino acid derivative called BPA, boronophenylalanine) will capture the neutrons. As a result from the neutron capture the boron atoms will split into two, producing helium and lithium ions. The helium and lithium ions, in turn, have only a short pathlength in tissue (about 5 micrometers) and will deposit their cell damaging effect mainly within the tumor provided that the boron carrier (BPA) has accumulated in the tumor. In practice, the study participants will receive BPA as an approximately 2-hour intravenous infusion, following which the tumor is irradiated with low energy (epithermal) neutrons obtained from a nuclear reactor at the BNCT facility. BNCT requires careful radiation dose planning, but neutron irradiation will last approximately only for one hour. In this study BNCT will be repeated, and the 2 treatments will be given 3 to 5 weeks apart. The study hypothesis is that head and neck cancers that have recurred following conventional radiotherapy might accumulate the boron carrier compound, and might respond to BNCT.

DETAILED DESCRIPTION:
This is a single BNCT-facility, non-randomized, non-comparative, open-label, phase I to II trial to determine the value of BNCT in the treatment of inoperable, irradiated, locally advanced cancers of the head and neck region. An attempt to perform 18F-labeled boronophenylalanine (18F-BPA) SPECT or PET imaging will be made before BNCT. Patients whose tumor uptake is >2.5 times that of the corresponding normal head and neck tissue will be enrolled, and treated with a single fraction BPA-based BNCT twice, 3 to 5 weeks apart. Another 18F-BPA SPECT or PET study may be performed 1 to 3 months after BNCT to determine the SPECT/PET response.

The neutron irradiation site is the FiR 1 reactor site, located at Otaniemi, Espoo, Finland, about 6 kilometers from the Helsinki University Central Hospital, Helsinki, where patient evaluation and post-irradiation care will take place.

Prior to BNCT, BPA is infused as a fructose complex (l-BPA-F) into a peripheral vein over 2 hours. Blood samples will be taken for monitoring whole blood boron concentration before starting the BPA infusion, and thereafter at 20 to 40 minute intervals during the infusion, following infusion, and after delivering neutron irradiation. The blood samples will be analyzed for blood boron concentration to estimate the average blood boron concentration during neutron irradiation.

All patients will be evaluated for response using CT or magnetic resonance imaging (MRI).

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed, malignant head and neck cancer.
* Inoperable tumor, prior surgery may or may not have been done.
* Prior radiotherapy or chemoradiotherapy has been given.
* If prior SPECT or PET with 18F-BFA has been done, BPA needs to accumulate at least 2.5 times more in the tumor than in the corresponding contralateral normal tissue.
* WHO performance status <3.
* WBC >2,500/mm3, platelets >75,000/mm3, serum creatinine <180 umol/L.
* A written informed consent.

Exclusion Criteria:

* Lymphoma or other tumor type that is expected to respond to cancer chemotherapy or to a dose of conventional radiation therapy that can be safely given.
* A non-experimental, effective treatment option is available.
* Expected survival less than 3 months.
* Concomitant systemic chemotherapy (prior cancer chemotherapy is allowed).
* Other concurrent experimental therapy, or such therapy is being planned to be given.
* Less than 3 months since prior radiation therapy.
* Untreated or severe, treated congestive heart failure or renal failure.
* A cardiac pace-maker or an unremovable metal implant present in the head and neck region that will interfere with MRI-based dose-planning.
* Restlessness or inability to lie in a cast for 30 to 60 minutes.
* Clinical follow-up after therapy cannot be arranged or the patient is not willing to participate in follow-up.
* Pregnancy.
* Age less than 18.
* The patient is not able to understand the treatment options.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2003-12; Primary Completion 2008-10 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
treatment response | 1 year

SECONDARY OUTCOMES:
time to progression | 2 years
safety | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Heikki T Joensuu, M.D., prof., Principal Investigator — Helsinki University Central Hospital
Locations (1):
- Department of Oncology, Helsinki University Central Hospital, Helsinki, Finland

REFERENCES:
- [Background] Kouri M, Kankaanranta L, Seppala T, Tervo L, Rasilainen M, Minn H, Eskola O, Vahatalo J, Paetau A, Savolainen S, Auterinen I, Jaaskelainen J, Joensuu H. Undifferentiated sinonasal carcinoma may respond to single-fraction boron neutron capture therapy. Radiother Oncol. 2004 Jul;72(1):83-5. doi: 10.1016/j.radonc.2004.03.016. PMID 15236879
- [Background] Joensuu H, Kankaanranta L, Seppala T, Auterinen I, Kallio M, Kulvik M, Laakso J, Vahatalo J, Kortesniemi M, Kotiluoto P, Seren T, Karila J, Brander A, Jarviluoma E, Ryynanen P, Paetau A, Ruokonen I, Minn H, Tenhunen M, Jaaskelainen J, Farkkila M, Savolainen S. Boron neutron capture therapy of brain tumors: clinical trials at the finnish facility using boronophenylalanine. J Neurooncol. 2003 Mar-Apr;62(1-2):123-34. doi: 10.1007/BF02699939. PMID 12749708
- [Derived] Porra L, Wendland L, Seppala T, Koivunoro H, Revitzer H, Tervonen J, Kankaanranta L, Anttonen A, Tenhunen M, Joensuu H. From Nuclear Reactor-Based to Proton Accelerator-Based Therapy: The Finnish Boron Neutron Capture Therapy Experience. Cancer Biother Radiopharm. 2023 Apr;38(3):184-191. doi: 10.1089/cbr.2022.0059. Epub 2022 Oct 21. PMID 36269660
- [Derived] Kankaanranta L, Seppala T, Koivunoro H, Saarilahti K, Atula T, Collan J, Salli E, Kortesniemi M, Uusi-Simola J, Valimaki P, Makitie A, Seppanen M, Minn H, Revitzer H, Kouri M, Kotiluoto P, Seren T, Auterinen I, Savolainen S, Joensuu H. Boron neutron capture therapy in the treatment of locally recurred head-and-neck cancer: final analysis of a phase I/II trial. Int J Radiat Oncol Biol Phys. 2012 Jan 1;82(1):e67-75. doi: 10.1016/j.ijrobp.2010.09.057. Epub 2011 Feb 6. PMID 21300462